CLINICAL TRIAL: NCT00370656
Title: A Double-blind, Randomised, Parallel Groups Investigation Into the Effects of Pregabalin, Duloxetine and Amitriptyline on Aspects of Pain, Sleep, and Next Day Performance in Patients Suffering From Diabetic Peripheral Neuropathy
Brief Title: Effects of Pregabalin, Duloxetine & Amitriptyline on Pain & Sleep
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Professor Anthony Nicholson, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRC 235
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathies
Keywords: Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases | interventions — Pregabalin; Duloxetine Hydrochloride; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Pregabalin — capsule, 150mg bd, 300mg bd
Drug: Duloxetine — Capsule, 60mg on, 60mg bd
Drug: Amitriptyline — Capsule. 25 mg bd, 25 mg om and 50 mg on

SUMMARY:
The purpose of this study is to assess the effectiveness of pregabalin, duloxetine and amitriptyline compared with placebo in reducing pain in diabetic patients as assessed by Brief Pain Inventory (BPI).

DETAILED DESCRIPTION:
Little is understood concerning the interaction of pain with sleep. Pain may disrupt sleep leading to daytime sleepiness and poor sleep can increase the perception of pain. There is uncertainty concerning the most effective way in which medication could be used to ease pain and poor sleep in patients such as those with diabetic peripheral neuropathy. Various drugs have been tried or proposed, and these include amitriptyline, pregabalin and duloxetine.

Amitriptyline is believed to relieve pain and improve sleep, though there is little evidence of its beneficial effects on sleep. Furthermore, even at low doses, it affects reaction time, attention, memory, information processing.

In two studies with duloxetine, it has been shown to significantly reduce pain compared with placebo, although little data are available on the usefulness of this compound in the management of pain with poor sleep.

Pregabalin has been shown to be effective in reducing pain, and therefore improving sleep. It has also been demonstrated that it has limited potential to affect daytime cognition. In another study gabapentin (a compound structurally related to pregabalin) demonstrated superior efficacy in the management of pain compared to amitriptyline.

Therefore this study will assess the effectiveness of pregabalin, duloxetine and amitriptyline compared with placebo in reducing pain associated with diabetes and poor sleep.

As the incidence of diabetes is predicted to increase in future years and as a consequence so will the cases of diabetic peripheral neuropathy (DPN), this research will serve to provide essential information on sleep and DPN which will be beneficial now and in the future.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or above
2. Have a diagnosis of Diabetes mellitus for at least a year
3. Agree not to smoke whilst resident in the CRC
4. Able to understand the patient information sheet and provide written informed consent
5. Score above 12 on the LANSS
6. Have neuropathic pain of diabetic origin
7. Score above 25 on MMSE
8. Willing to withdraw, under the guidance of their diabetologist, from any current pain medication prior to their first visit to the sleep laboratory. Duration of withdrawal will be at least equivalent to 5 half-lives and will be of a relevant duration given the particular medication used.

Exclusion Criteria:

1. There is evidence of an end stage disease of a major system (hepatic, renal, respiratory, haematologic (PA), immunologic, cardiovascular, inflammatory, rheumatology, active infections, peripheral vascular disease, untreated endocrine(hypothyroid)
2. There is evidence of a recent ischaemic event
3. There is evidence of recurrent and/or severe hypoglycemia requiring assistance in last 3 years
4. Evidence of sleep pathology that would interfere with the assessment of treatment (assessed on habituation night)
5. Currently receiving treatment for malignancy
6. Suffer from seizures including epilepsy
7. There is evidence of a history of dependence on or abuse of alcohol/recreational drugs
8. Need to use a wheel chair (incompatible with studies in a sleep laboratory)
9. Involved in a clinical trial in last 3 months
10. Pregnant, lactating or inadequate contraception
11. Vision inadequate for the performance tests (as assessed at screening)
12. Colour Blind
13. Will not co-operate with study procedures
14. Will not give permission to inform GP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Whether there is a reduction in subjective pain as assessed by the Brief Pain Inventory. | December 2008

SECONDARY OUTCOMES:
Whether there has been an improvement in sleep continuity and subjective sleep, morning after cognitive and psychomotor performance, and quality of life (QoL). | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Professor AN Nicholson, Principal Investigator — University of Surrey; Dr D Kerr, Principal Investigator — Royal Bournemouth Hospital; Dr D Coppini, Principal Investigator — Poole General Hospital
Locations (3):
- United Kingdom (3):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Poole General Hospital, Poole, Dorset
  - University of Surrey Clinical Research Centre, Guildford, Surrey

REFERENCES:
- [Derived] Boyle J, Eriksson ME, Gribble L, Gouni R, Johnsen S, Coppini DV, Kerr D. Randomized, placebo-controlled comparison of amitriptyline, duloxetine, and pregabalin in patients with chronic diabetic peripheral neuropathic pain: impact on pain, polysomnographic sleep, daytime functioning, and quality of life. Diabetes Care. 2012 Dec;35(12):2451-8. doi: 10.2337/dc12-0656. Epub 2012 Sep 18. PMID 22991449